CLINICAL TRIAL: NCT06365983
Title: Comparison of Free Gingival Graft and Linear Incision Techniques to Obtain Connective Tissue Graft in the Treatment of Multiple Gingival Recessions: a 12-month Non-inferiority Randomized Trial
Brief Title: Comparison of Free Gingival Graft and Linear Incision for Connective Tissue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alex Nogueira Haas, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRGS-Cassio
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Connective Tissue; Gingiva; Gingival Recession; Humans
Keywords: Free Gingival Graft; Linear Technique; Root Coverage
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: A randomized controlled non-inferiority trial will be conducted with 24 individuals aged 18 or older, who are periodontally healthy and require root coverage in bilateral multiple RT1-type recessions involving at least two teeth on each side of the mouth. The number of teeth to be covered must be equal on both sides to avoid imbalance in patient-centered comparisons.
Who Masked: Outcomes Assessor
Masking Description: All sample randomization procedures will be carried out by a researcher not involved in treatments and clinical examinations. An external researcher not affiliated with the study will be responsible for maintaining participant allocation confidentiality. Sides will be identified by numbers stored in opaque, sealed envelopes with the randomization sequence. Outcome assessors will be blinded to the experimental group to which participants belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Gingival Graft (Active Comparator)
  Interventions: Procedure: Connective Tissue with Free Gingival Graft
- Linear Incision (Experimental)
  Interventions: Procedure: Connective Tissue with Linear Incision

INTERVENTIONS:
Procedure: Connective Tissue with Free Gingival Graft — The de-epithelialized free gingival grafting will begin with two horizontal incisions, 1.0 to 1.5 mm apical to the margin of the soft tissue of the adjacent teeth and two vertical incisions to delimit the area to be grafted. Along the coronal horizontal incision, the blade will be oriented almost perpendicular to the bone surface, and once an adequate thickness of soft tissue is obtained, it will be rotated to become almost parallel to the external surface of the palate. The graft thickness will be maintained uniform and the wound will be protected with absorbable collagen sponge derived from swine (Spongostan; Ethicon, Somerville, USA) and maintained with compressive sutures with non-absorbable 5-0 monofilament thread (Microsuture, São Paulo), anchored to the soft tissue apical to the area of the palatal wound. Immediately after suture completion, drops of high viscosity cyanoacrylate adhesive (PeriAcryl 90 HV; Glustitch, Delta, Canada) will be applied.
  Arms: Free Gingival Graft
Procedure: Connective Tissue with Linear Incision — The linear technique (Lorenzana ER, Allen EP 2000) will begin with a horizontal incision 2 mm apical to the gingival margin, perpendicular to the palate, which is deepened to the bone crest. Next, a second incision is made to divide the flap and expose the connective tissue bed. The thickness of the outer portion of the flap should be at least 1 mm, with uniformity throughout its extension to reduce the risk of epithelial tissue necrosis. Subsequently, internal lateral incisions (mesial and distal) and the base incision will be made, connecting the vertical incisions to delineate horizontal and vertical boundaries. Immediately after graft removal, an absorbable hemostatic collagen sponge derived from swine (Spongostan; Ethicon, Somerville, USA) will be placed and sutured using non-absorbable 5-0 monofilament thread (Microsuture, São Paulo).Immediately after suturing is completed, drops of high viscosity cyanoacrylate adhesive (PeriAcryl 90 HV; Glustitch, Delta, Canada) will be applied.
  Arms: Linear Incision

SUMMARY:
A randomized controlled non-inferiority trial will be conducted with 24 individuals aged 18 or older, who are periodontally healthy and require root coverage in bilateral multiple RT1-type recessions involving at least two teeth on each side of the mouth. The number of teeth to be covered must be equal on both sides to avoid imbalance in patient-centered comparisons.

Patients included in the study will undergo the bilateral multiple root coverage technique with coronally repositioned flap (Zucchelli and De Sanctis) in both groups. The donor areas for connective tissue will be the hard palate region, with grafts harvested using the linear technique on one side and the free de-epithelialized gingival graft technique on the other side.

Each patient will undergo a preparatory phase for study inclusion, consisting of supragingival scaling, polishing, and oral hygiene instructions at least 3 weeks before study inclusion. Patients will be instructed on personalized and proper use of toothbrush, dental floss, and/or interdental brush.

All surgical procedures in both groups will be performed by the same operator (CCO). Randomization will determine the side to be operated on first. The other side will be operated on after 30 days or until the patient reports complete absence of symptoms in the area of the first surgery to avoid confusion in patient-centered outcomes regarding pain and satisfaction with the techniques.

Outcomes evaluated at 3, 6, 9, and 12 months include: gingival recession depth, probing depth, visible plaque, bleeding on probing, width of keratinized tissue, three-dimensional tissue assessment from intraoral scanning, and quality of life related. Linear and logistic generalized estimating equation models considering the longitudinal nature of the study will be used for data analysis.

INCLUSION CRITERIA Patients aged 18 or older requiring root coverage in bilateral multiple recessions involving at least two teeth on each side of the mouth will be included. The number of teeth to be covered must be equal on both sides to avoid imbalance in patient-centered comparisons. Recessions should be RT1 type according to the 2017 Workshop on the Classification of Periodontal Conditions and Diseases (Jepsen et al. 2018) and without non-carious cervical lesions.

EXCLUSION CRITERIA

Individuals will not be considered eligible if they:

* Present any form of immunological compromise;
* Have diseases or systemic conditions contraindicating surgical procedures or affecting periodontal healing pattern, such as diabetes and autoimmune diseases;
* Present active periodontitis, defined by presence of >=10% subgingival bleeding and probing depth and clinical attachment loss proximal >4mm (Tonetti et al. 2018);
* Are current or ex-smokers;
* Have allergies to ibuprofen and chlorhexidine digluconate.

Research Objective:

PRIMARY OBJECTIVE The overall objective of this study is to compare free gingival graft and subepithelial connective tissue graft in outcomes related to multiple recession coverage.

SECONDARY OBJECTIVE

Compare the two grafts in terms of clinical outcomes of root coverage; Compare the two grafts in terms of digital outcomes of root coverage obtained in scanning and tomography; Compare the two grafts in terms of patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 or older requiring root coverage in bilateral multiple recessions involving at least two teeth on each side of the mouth will be included. The number of teeth to be covered must be equal on both sides to avoid imbalance in patient-centered comparisons. Recessions should be RT1 type according to the 2017 Workshop on the Classification of Periodontal Conditions and Diseases (Jepsen et al. 2018) and without non-carious cervical lesions.

Exclusion Criteria:

Individuals will not be considered eligible if they:

* Present any form of immunological compromise;
* Have diseases or systemic conditions contraindicating surgical procedures or affecting periodontal healing pattern, such as diabetes and autoimmune diseases;
* Present active periodontitis, defined by presence of >=10% subgingival bleeding and probing depth and clinical attachment loss proximal >4mm (Tonetti et al. 2018);
* Are current or ex-smokers;
* Have allergies to ibuprofen and chlorhexidine digluconate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of root coverage | 12 months
  Final minus baseline recession depth divided by baseline value

SECONDARY OUTCOMES:
Recession depth | Baseline, 3, 6, 9 e 12 months
  Measurement from the cementoenamel junction to the most apical extension of the gingival margin

CONTACTS AND LOCATIONS:
Locations (1):
- Alex Nogueira Haas, Porto Alegre, Rio Grande do Sul, Brazil